CLINICAL TRIAL: NCT01750749
Title: Autologous Bone Marrow Derived Cells in the Treatment of Venous Leg Ulcers Pilot Study
Brief Title: Cell Therapy for Venous Leg Ulcers Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital de Clínicas Dr. Manuel Quintela (Other)
Responsible Party: Principal Investigator, Cristina Touriño, MD, PhD, Coordinator of the, Hospital de Clínicas Dr. Manuel Quintela
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUV2011
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Venous Ulcer
Keywords: Venous ulcer; Cell therapy
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous BMDC implantation at the venous ulcer (Experimental): Autologous BMDC implantation at the venous ulcer in conjunction with SOC treatment (advanced wound management plus pressure therapy)
  Interventions: Biological: Autologous BMDC implantation at the venous ulcer

INTERVENTIONS:
Biological: Autologous BMDC implantation at the venous ulcer — An autologous bone marrow derived cell concentrate is obtained by bone marrow harvest (300 ml) from the iliac crest and subsequent processing using 6% hydroxyethyl starch to concentrate nucleated cells. The cells are injected using a 27 Gauge needle, in aliquots of 0.2 ml, along the venous ulcer edge. SOC treatment consisting of advanced wound management plus pressure therapy is administered simultaneously.

SUMMARY:
Chronic venous leg ulcers (CVU) represent a medical problem associated with significant morbidity, increased work absenteeism and earlier retirement as a consequence of disability. This strongly affects the patient's quality of life and has a significant economic impact on healthcare systems.

Reports of studies with animal models show that treatment with bone marrow-derived stem cells has a beneficial effect in healing chronic skin wounds.

The purpose of this pilot study is to determine the safety and feasibility of cell therapy with bone marrow derived cells (BMDC) as a complementary healing therapy in chronic venous leg ulcers, and in addition to evaluate its effectiveness. The knowledge gained in the pilot study will be used to refine the clinical protocol procedures of a subsequent randomized study.

Patients with venous legs ulcers meeting eligibility criteria and providing appropriate written informed consent will be enrolled for study participation. Enrolled patients will receive Autologous BMDC implantation at de venous ulcer in conjunction with standard of care (SOC) treatment.

During follow up, adverse events will be assessed by ulcer clinical examination. Effectiveness of the experimental treatment will be assessed by evaluating ulcer healing (reduction of the ulcer area) and pain reduction over a six-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 75 years
* Patients with primary venous insufficiency
* Patients with venous ulcers with area larger than 2 cm2, who have received SOC treatment in the previous three months.
* Ulcers with negative bacterial cultures or with polymicrobial flora.

Exclusion Criteria:

* Patients with decompensated heart failure.
* Patients with lower limb edema of nonvenous etiology.
* Patients with diagnosis of diabetes mellitus.
* Patients with body mass index (BMI) ≤ 18.5 or > 40.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Reduction of the ulcer area at 2 months | 2 months
  Measurement of the ulcer area (cm2) and comparison with baseline.
Reduction of the ulcer area at 4 months | 4 months
  Measurement of the ulcer area (cm2) and comparison with baseline.
Reduction of the ulcer area at 6 months | 6 months
  Measurement of the ulcer area (cm2) and comparison with baseline.

SECONDARY OUTCOMES:
Pain reduction at 2 months | 2 months after intervention
  Assess of pain by visual analog score
Pain reduction at 4 months | 4 months after intervention
  Assess of pain by visual analog score
Pain reduction at 6 months | 6 months after intervention
  Assess of pain by visual analog score
Absence of adverse events related with the intervention | From date of cells implantation until the date of the event, assesed up to 7 days
  Clinical examination of the site of cells implantation for signs of infection, hematoma, edema or eczema. Asses of pain by visual analog score.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Otero, MD, Principal Investigator — Cátedra de Dermatología; Cristina Touriño, MD, PhD, Study Director — Área de Terapia Celular y Medicina Regenerativa
Locations (1):
- Universidad de la República- Hospital de Clínicas Dr. Manuel Quintela, Montevideo, Uruguay